CLINICAL TRIAL: NCT03440281
Title: Maternal Serum Homocysteine Levels and Uterine Artery Pulsatility Index as Predictors of Spontaneous Preterm Labor
Brief Title: Maternal Serum Homocysteine Levels and Uterine Artery Pulsatility Indices in Preterm Labor
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Walid Anwar Murad, Assisstant proffessor of Obestetrics &Gynecology, Benha University
Other Study IDs: 1182015
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm group: included pregnant females delivered prior to completed 37 weeks of gestation. All participants underwent assessment of uterine artery Doppler indices and maternal serum homocysteine estimation
  Interventions: Diagnostic Test: Uterine artery doppler; Diagnostic Test: Maternal serum homocysteine estimation
- Term group: Included pregnant females delivered after completed 37 weeks of gestation. All participants underwent assessment of uterine artery Doppler indices and maternal serum homocysteine estimation
  Interventions: Diagnostic Test: Uterine artery doppler; Diagnostic Test: Maternal serum homocysteine estimation

INTERVENTIONS:
Diagnostic Test: Uterine artery doppler — Uterine artery Doppler pulsatility indices
Diagnostic Test: Maternal serum homocysteine estimation

SUMMARY:
Study included all pregnant women admitted with threatened preterm labor during the study period. All participants underwent estimation of maternal serum homocysteine level and assessment of uterine artery Doppler indices.

DETAILED DESCRIPTION:
Prospective cohort study. Study approval by local ethics committee. Informed written consent. Study included all pregnant women admitted with threatened preterm labor during the study period. All participants underwent estimation of maternal serum homocysteine level and assessment of uterine artery Doppler indices.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* More than 28 and less than 35 gestational weeks.
* Threatened preterm labor

Exclusion Criteria:

* Medical disorders complicating pregnancy
* Obstetric conditions complicating pregnancy (e.g., placenta previa, multiple gestation,PPROM, ....etc)
* Fetal anomalies or distress

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant with singleton pregnancy, more than 28 and less than 35 gestational weeks.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
The accuracy of serum homocysteine levels and uterine artery pulsatility indices (UtA-PI ) for prediction of preterm labor | Single measurement at the end of the study ( around 37 gestational weeks)
  Sensitivity (%), specificity (%), positive predictive value (%), negative predictive value (%), positive likelihood ratio (number), negative likelihood ratio (number), accuracy (%) of serum homocysteine and UtA-PI for prediction of preterm labor

SECONDARY OUTCOMES:
Gestational age at delivery | Single measurement at the end of the study ( around 37 gestational weeks)
  Gestational age at delivery (Weeks),
Demographic and clinical characteristics of the study groups | Single measurement on the day one of hospital admission between 28-35 gestational weeks
  Maternal age (year), Body mass index (kilogram per squared meter), Gestational age at admission (Weeks), Maternal serum Homocysteine level ( micromoles/liter), uterine artery pulsatility index ( number)

IPD SHARING:
Plan to Share IPD: No